CLINICAL TRIAL: NCT05381454
Title: An Open Label Study in Adults to Test the Efficacy of Mitoquinone/Mitoquinol Mesylate as Prophylaxis for Development of Severe Viral Illness
Brief Title: An Open Label Study in Adults to Test the Efficacy of Mitoquinone/Mitoquinol Mesylate to Prevent Severe Viral Illness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Theodoros Kelesidis, MD, PhD, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-21-1940
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Viral Infection; Antiviral Treatment; COVID-19
Keywords: Respiratory Viral Infection; Antiviral treatment; COVID-19; Prophylaxis COVID-19
MeSH Terms: conditions — COVID-19 | interventions — mitoquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MitoQ (Experimental): Treatment group
  Interventions: Drug: Mitoquinone/mitoquinol mesylate
- Control group (No Intervention): Control group

INTERVENTIONS:
Drug: Mitoquinone/mitoquinol mesylate — Mitoquinone/mitoquinol mesylate
  Other Names: MitoQ
  Arms: MitoQ

SUMMARY:
Open label clinical trial of persons (adults) that will determine the safety and efficacy of the diet supplement oral mitoquinone/mitoquinol mesylate (Mito-MES) to prevent the development and progression of severe viral infections like COVID-19 after high-risk exposure to a person with possible respiratory viral infection such as SARS-CoV-2 infection in persons who will receive Mito-MES compared to persons who will not receive Mito-MES (controls).

DETAILED DESCRIPTION:
Overview of study design Open label clinical trial of persons (adults) that will determine the safety and efficacy of the diet supplement oral mitoquinone/mitoquinol mesylate (Mito-MES) to prevent the development and progression of severe viral infections like COVID-19 after high-risk exposure to a person with possible respiratory viral infection such as SARS-CoV-2 infection in persons who will receive Mito-MES compared to persons who will not receive Mito-MES (controls). A study participant will have the option to enroll either in the treatment arm or the control arm (no intervention but will complete relevant questionnaires and study procedures).

Efficacy: To determine the efficacy of the treatment with mito-MES 20 mg daily for up to 14 days compared to no treatment with mito-MES to prevent development of severe clinical symptoms of any viral infection in high-risk close household contacts of cases with viral infection. Viral infection will be defined clinically based on history obtained by the investigator who is an infectious diseases physician and stringent criteria will be followed. Viral infection will be defined as presence of at least two new onset independent symptoms or signs (fever) of respiratory disease that cannot be attributed to bacterial cause (for example the combination of runny nose and sore throat is very characteristic of a viral illness). The combination of fever and cough is not specific enough presentation since it can be attributed also to bacterial bronchitis or pneumonia. A study participant with chronic allergies or chronic sinusitis or asthma will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled participants must meet the following criteria:

  * Age 18-65 years old.
  * Asymptomatic (no symptoms of viral infection) on study entry.
  * Exposure to a person with at least two new onset independent symptoms or signs (fever) of respiratory viral disease
  * High risk exposure without use of masks and physical distancing to suspected case of viral illness (based on established symptoms of viral illness) in the household within 3 days prior to study entry. Rationale: Antivirals are most efficacious when given as early as possible post exposure.
  * Ineligible for FDA approved alternative treatments to prevent progression to severe COVID-19 based on established criteria https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/people-with-medical-conditions.html or FDA approved alternative treatment cannot be obtained or not indicated (e.g. allergy).
  * Without established significant coronary artery/vascular disease, lung, stroke, kidney, liver, heart disease) based on history.
  * Adequate renal function. This is defined as absence of documented history of any kidney disease.

Exclusion Criteria:

* Participants who meet any of the following criteria at screening will be excluded from the study:

  1. Use of Coenzyme Q10 or Vitamin E < 120 days from enrollment
  2. Women with variations in physiological functions due to hormones that may effect immune function and (taking hormones, pregnant, breastfeeding, on contraceptives).
  3. Pregnant (based on history).
  4. History of known gastrointestinal disease (such as gastroparesis) that may predispose patients to nausea. Gastrointestinal symptoms are the most common side effects of MitoQ.
  5. History of auto-immune diseases
  6. Chronic viral hepatitis
  7. History of underlying cardiac arrhythmia
  8. History of severe recent cardiac or pulmonary event
  9. A history of a hypersensitivity reaction to any components of the study drug or structurally similar compounds including Coenzyme Q10 and idebenone
  10. Unable to swallow tablets
  11. Use of any investigational products within 28 days of study enrollment
  12. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease
  13. Participants who are eligible for FDA approved alternative treatments to prevent progression to severe COVID-19 based on established criteria https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/people-with-medical-conditions.html

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Kelesidis, MD PHD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Derived] Chen K, Jackson NJ, Kelesidis T. Mitoquinone mesylate as post-exposure prophylaxis against SARS-CoV-2 infection in humans: an exploratory single center pragmatic open label non-randomized pilot clinical trial with matched controls. EBioMedicine. 2024 Apr;102:105042. doi: 10.1016/j.ebiom.2024.105042. Epub 2024 Mar 11. PMID 38471990

RESULTS

PARTICIPANT FLOW:
Groups:
- MitoQ 20 mg orally daily: Treatment group
  Mitoquinone/mitoquinol mesylate: Mitoquinone/mitoquinol mesylate
- Control: Control group
Period: Overall Study
Arm/Group | MitoQ 20 mg orally daily | Control
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: General population
Groups:
- Total: Total of all reporting groups
Arm/Group | MitoQ 20 mg Orally Daily | Control | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.5 [34.8 to 42] | 44.0 [42.0 to 46] | 41.5 [37.3 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 17 | 21 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 37 | 38 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Vaccinated with COVID-19 mRNA vaccine within 6 months prior to exposure [Count of Participants; unit: Participants] | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Illness
Description: Development of viral illness based on diagnostic test
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitoQ 20 mg orally daily | Control
Number analyzed (Participants) | 40 | 40
Participants | 12 | 30

2. Primary Outcome: Severity Score of Symptoms of Viral Illness
Description: Severity of viral illness based on a quantitative score system. Each of the above 14 symptoms will be given a score based on severity: 1 for mild, 2 for moderate, 3 for severe. Then a total severity score will be estimated (range of score is 0-42). Common example: a person with mild coryza, sore throat and cough will be given a score of 3. A higher score means worse outcome
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MitoQ 20 mg orally daily | Control
Number analyzed (Participants) | 40 | 40
score on a scale | 2.0 [1.75 to 2.25] | 3.0 [2.5 to 4.5]

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events as Assessed by the Proportion of Participants Exhibiting Adverse Events of Any Grade
Description: Assessment of adverse events up to 14 days post initiation of therapy. Adverse events: the proportion of participants exhibiting adverse events of any grade
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitoQ 20 mg orally daily | Control
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Fever
Description: Development of new onset fever (T> 100.3 F or 38C) based on documented
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitoQ 20 mg orally daily | Control
Number analyzed (Participants) | 40 | 40
Participants | 0 | 10

5. Secondary Outcome: Number of Participants With Any Symptoms of Viral Illness
Description: Duration in days of at least three respiratory/systemic symptom of viral illness. This means that if any of the listed symptoms last more than a day, then the participant is considered to have a viral illness. (Symptom 1: fever, Symptom 2: cough, Symptom 3: coryza, Symptom 4: sore throat, Symptom 5: shortness of breath, Symptom 6: chills, Symptom 7: fatigue, Symptom 8: loss of smell or taste, Symptom 9: myalgias, Symptom 10: arthralgias, Symptom 11: headache, Symptom 12: nausea, Symptom 13: vomiting, Symptom 14: diarrhea
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitoQ 20 mg orally daily | Control
Number analyzed (Participants) | 40 | 40
Participants | 4 | 23

ADVERSE EVENTS:
Time Frame: 14 days
Description: As per clinicaltrials.gov definitions. Zero means that all study participants were observed for adverse events and none was observed. The Total Number of Participants at Risk equals the number of participants Started in the Participant Flow module.
Arm/Group | MitoQ 20 Mg orally daily | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT05381454/Prot_SAP_000.pdf